CLINICAL TRIAL: NCT06246253
Title: Bone Formed Labial to the Implant in Relation to the Horizontal Gap Dimension in Immediate Implant Placement. A CBCT Study
Brief Title: Socket Evaluation System to Predict Labial Bone Formation Around Immediate Implants. A Retrospective Cone Beam Computed Tomography Analysis.
Status: Completed | Type: Observational
Sponsor: Misr International University (Other)
Collaborators: International Dental Contiuing Education (Network)
Responsible Party: Principal Investigator, Ahmed Abo El Futtouh, Owner & Comprehensive Implant Training Program Director, International Dental Contiuing Education
Other Study IDs: IDCE-12207025
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2022-01

CONDITIONS: Immediate Implant Placement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Virtual implant placement following safe angle concept
  Interventions: Procedure: Virtual implant placement following safe angle concept
- actual implant placement following safe angle concept
  Interventions: Procedure: actual implant placement following safe angle concept

INTERVENTIONS:
Procedure: Virtual implant placement following safe angle concept — Virtual implant placement following safe angle concept in anterior maxillary teeth.
  Groups: Virtual implant placement following safe angle concept
Procedure: actual implant placement following safe angle concept — actual implant placement following safe angle concept in anterior maxillary teeth
  Groups: actual implant placement following safe angle concept

SUMMARY:
Palate implant placement in extraction sockets, with a minimum of 2 mm between the implant and the inner side of the facial socket wall, has been advised as a step towards a 3D restorative-driven posture. The buccal gap left by this palatal location is identified by the term "jumping gap" or "jumping distance," which describes the capacity of bone to fill the void and bridge the horizontal gap. The gap is made up of a vertical and horizontal component. Significantly, this gap denotes the future buccal bone that will directly contribute to the buccal contour and impact the soft tissue levels, thus influencing the implant's final appearance. Consequently, it is now considered desirable to have a bigger horizontal gap since more newly created buccal bone is predicted to occur in areas with larger horizontal gaps.

ELIGIBILITY:
Inclusion Criteria:

* anterior maxillary teeth
* Immediate implant placement

Exclusion Criteria:

* fractured apical part of the root
* teeth with apical resorption or displacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Immediate implant placement in anterior maxillary teeth
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
labial gap dimension | pre and immediately after implant placement
  labial gap dimension will be measured as an area from the preoperative and immediatly post operative CBCTs

CONTACTS AND LOCATIONS:
Locations (1):
- International Dental Continuing Education (IDCE) centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No